CLINICAL TRIAL: NCT07095361
Title: Once Daily Intrapleural Enzyme Therapy in Complicated Parapneumonic Effusion or Empyema (ONLY ONCE)
Brief Title: Once Daily Intrapleural Enzyme Therapy in Complicated Parapneumonic Effusion or Empyema
Acronym: ONLY ONCE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-1309
Record Dates: First submitted 2025-07-11; First posted 2025-07-31 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Pleural Infection Bacterial; Pleural Infections; Pleural Infections and Inflammations; Empyema, Pleural; Empyema; Complicated Pleural Effusion/ Empyema; Pleural Effusion Associated With Pulmonary Infection; Pleural Effusion
Keywords: Lytics; Intrapleural enzyme therapy; Once daily; lytic therapy
MeSH Terms: conditions — Inflammation; Empyema, Pleural; Empyema; Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Once daily intrapleural enzyme therapy (Experimental): Participants will receive intrapleural enzyme therapy (IET) once daily for 3 consecutive days.
  Interventions: Drug: Fibrinolytic once daily; Drug: DNA degradation once daily
- Twice daily intrapleural enzyme therapy (Active Comparator): Participants will receive intrapleural enzyme therapy (IET) twice daily for 3 consecutive days.
  Interventions: Drug: Fibrinolytic twice daily; Drug: DNA degradation twice daily

INTERVENTIONS:
Drug: Fibrinolytic once daily — tissue plasminogen activator (tPA) 10mg will be administered once a day as part of intrapleural enzyme therapy (IET) for 3 consecutive days.
  Other Names: once daily lytics; tPA once daily
  Arms: Once daily intrapleural enzyme therapy
Drug: Fibrinolytic twice daily — tissue plasminogen activator (tPA) 10mg will be administered twice a day as intrapleural enzyme therapy for 3 consecutive days.
  Other Names: lytics twice daily; tPA twice daily
  Arms: Twice daily intrapleural enzyme therapy
Drug: DNA degradation once daily — Deoxyribonuclease (DNase) 5mg will be administered once a day as intrapleural enzyme therapy (IET) for 3 consecutive days.
  Other Names: DNase once daily; lytics once daily
  Arms: Once daily intrapleural enzyme therapy
Drug: DNA degradation twice daily — Deoxyribonuclease (DNase) 5mg will be administered twice a day as intrapleural enzyme therapy for 3 consecutive days.
  Other Names: lytics twice daily; DNase twice daily
  Arms: Twice daily intrapleural enzyme therapy

SUMMARY:
The goal of this clinical trial is to find out if giving certain medications once a day works just as well as giving them twice a day to treat infections around the lungs (called pleural infections). These medications-tissue plasminogen activator (tPA) and deoxyribonuclease (DNase)-are placed through a chest tube into the space between the lung and the chest wall to help clear out the infection.

The investigators are trying to learn:

* Does using the medicine once a day work just as well as using it twice a day?
* Are there any differences in outcomes between patients who get the medicine once a day versus twice a day?
* Does more or less fluid remain in the chest (seen on a chest x-ray) depending on how often the medicine is given?

Participants will:

* Have an infection around their lung and will already be getting normal hospital care, including a chest tube to drain the infected fluid around their lung.
* Be asked to give permission to join the study.
* Be randomly chosen (like flipping a coin) to get the medications either once a day or twice a day through the chest tube.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from patient or patient's legally authorized representative (LAR) to participate in the study and HIPAA authorization for release of personal health information.
* Subject is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee.
* Age ≥ 18 years at the time of consent.
* Patient is admitted to the hospital and with a pleural effusion that is drained with a small-bore chest tube or one that allows for administration of IET
* Pleural fluid that is one of the following:

  (i) Macroscopically purulent or pleural fluid gram stain or culture positive for bacteria (ii) potential of hydrogen (pH) < 7.2 (iii) Pleural fluid glucose < 60mg/dL (iv) Pleural fluid Lactate Dehydrogenase (LDH) > 1,000 IU/L
* Patient is deemed a candidate to receive intrapleural enzyme therapy as defined by having a residual collection or persistent sepsis 24 hours after initial chest tube placement

Exclusion Criteria:

* Known pregnancy or lactating females
* Prisoners
* Age <18 years at time of consent
* Previous treatment with intra-pleural fibrinolytic agents, DNase, or both during the same hospital admission
* Known sensitivity or allergic reaction to DNAse or tPA
* Coincidental stroke, major hemorrhage (requiring blood transfusions within the last 5 days), major trauma, or major surgery within the last 5 days
* Previous pneumonectomy or active bronchopleural fistula on the affected side
* Therapeutic systemic anticoagulation or antiplatelet agents that cannot held for more than 48 hours prior to IET administration
* Expected survival of less than 3 months due to a pathologic condition other than that causing the pleural infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
IET Failure: Surgery and/or mortality at 90 days | 90 days
  Measure the rate of IET failure (defined as surgery and/or mortality at 90 days) in both once daily IET and twice daily IET groups.

SECONDARY OUTCOMES:
30 Day Mortality | 30 days
  Evaluate rate of mortality at 30 days between the participants receiving once daily IET and twice daily IET
Hospital length of stay | 90 days
  Evaluate length of hospitalization stay between the participants receiving once daily IET and twice daily IET
Oral Morphine Equivalents (OME) | From enrollment until day 3 of intervention
  Evaluate the difference in amount of oral morphine equivalents, which is a standardized method of reporting narcotic analgesic administration by converting opioid narcotics as determined by morphine milligram equivalents (MME) that would yield same result, for daily pain between once daily IET and twice daily IET.
Change of White Blood Cell Count | From enrollment until day 3 of intervention
  Evaluate the difference between white blood cell (WBC) count in units of cells per microliter (cells/μL) between once daily IET and twice daily IET.
Change in C-reactive Protein (CRP) level | From enrollment until day 3 of intervention
  Evaluate the difference between C-reactive protein (CRP) level, in milligrams per liter (mg/L) or milligrams per deciliter (mg/dL), between once daily IET and twice daily IET.
Change in Fever | From enrollment until day 3 of intervention
  Evaluate the difference between fever (in Celsius) between once daily IET and twice daily IET
Chest tube drainage amount | From enrollment until day 3 of intervention
  Evaluate the difference in amount (mL) of pleural fluid drained between once daily and twice daily IET groups
Duration of chest tube placement | 90 days
  Evaluate the number of days of chest tube placement between once daily and twice daily IET groups
Difference in pleural opacification on chest x-ray imaging between once daily IET and twice daily IET | From enrollment to 48 hours after completing 3 days of intrapleural enzyme therapy
  Measure the difference of pleural opacification on chest x-ray imaging, as measured in centimeter cubed (cm^3), between once daily IET compared to twice daily IET
Percent of participants who have pleural hemorrhage requiring blood transfusion | From enrollment to 48 hours after completing 3 days of intrapleural enzyme therapy
  Measure the percent of participants who have pleural hemorrhage requiring blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Jason Akulian, MD, MPH, Principal Investigator — University of North Carollina at Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with University of North Carolina (UNC).